CLINICAL TRIAL: NCT02366949
Title: An Open-label Randomized Two-arm Phase I Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of Oral BAY 1217389 in Combination With Weekly Intravenous Paclitaxel Given in an Intermittent Dosing Schedule in Subjects With Advanced Malignancies
Brief Title: Phase I Study of Oral BAY 1217389 in Combination With Intravenous Paclitaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17350; 2014-004821-41 (EudraCT Number)
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Medical Oncology
Keywords: Phase 1; Solid tumors; Breast cancer; Paclitaxel; MPS-1 inhibitor; Oncology
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Experimental Treatment (combination of BAY1217389 with paclitaxel in an intermittent dosing schedule) Expansion Cohort - Maximum tolerated dose of BAY1217389 and Paclitaxel
  Interventions: Drug: BAY1217389; Drug: Paclitaxel
- Arm 2 (Placebo Comparator): Standard Treatment (Single-agent Paclitaxel )
  Interventions: Drug: BAY1217389; Drug: Paclitaxel

INTERVENTIONS:
Drug: BAY1217389 — BAY1217389 will be given orally, with a starting dose of 0.25 mg twice daily, on D1, D2, D8, D9, D15 and D16 of a 28 day cycle. BAY1217389 will be dosed in combination with paclitaxel in Arm 1 (Experimental Treatment) and from Cycle 2 onwards in Arm 2 (Standard Treatment).
  After Maximum tolerated dose (MTD) has been defined, expansion cohorts will be conducted at the MTD dose of BAY1217389 and paclitaxel following an intermittent dosing schedule as defined in the dose escalation phase. Up to 12 to 15 breast cancer (triple negative) subjects are planned to be enrolled in the expansion cohort.
  In a higher dose level Cohort 4 > (or equal to) a relative bioavailability assessment of BAY1217389 liquid capsule formulation compared to BAY1217389 oral solution will be performed.
Drug: Paclitaxel — Paclitaxel will be given once per week IV at 90 mg/m^2 on D1, D8, and D15 of a 28 day cycle. Paclitaxel will be dosed as a single-agent in Cycle 1 of Arm 2 (Standard Treatment Arm), and in combination with BAY1217389 in Arm 1 (Experimental Treatment Arm) and from Cycle 2 onwards in Arm 2 (Standard Treatment Arm). After Maximum tolerated dose (MTD) has been defined, expansion cohorts will be conducted at the MTD dose of BAY1217389 and paclitaxel following an intermittent dosing schedule as defined in the dose escalation phase. Up to 12 to 15 breast cancer (triple negative) subjects are planned to be enrolled in the expansion cohort.

SUMMARY:
Determine the safety, tolerability, maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of oral BAY1217389 given in combination with intravenous (IV) paclitaxel using an intermittent dosing schedule (2 days on / 5 days off) in subjects with advanced malignancies.

DETAILED DESCRIPTION:
BAY1217389 is a potent and highly selective inhibitor of monopolar spindle 1 (MPS1) kinase activity. Human MPS1 is a serine threonine kinase, which functions as a core component of the spindle-assembly checkpoint (SAC), a key surveillance mechanism that monitors the attachment of spindle microtubules to the kinetochores of the chromosomes during pro-metaphase and halts the transitions to anaphase until all chromosomes are bi-oriented, fully attached, and correctly tensed at the metaphase plate. MPS1 is expressed in the mitosis phase of the cell cycle in proliferating cells. Overexpression of MPS1 has been observed in several cancer cell lines and tumor types, including lung and breast cancers.

Established anti-mitotic drugs such as vinca alkaloids, taxanes, or epothilones activate the SAC either by destabilizing or stabilizing spindle microtubules resulting in mitotic arrest. Prolonged arrest in mitosis forces a cell either into a mitotic exit without cytokinesis or into a mitotic catastrophe leading to cell death. In contrast, MPS1 inhibitors inactivate the SAC and accelerate progression of cells through mitosis eventually resulting in severe chromosomal missegregation, mitotic catastrophe, and cell death. Consequently, MPS1 inhibition leads to failure of cells to arrest in mitosis in response to anti-mitotic drugs. Thus, the combination of microtubule-interfering agents and MPS1 inhibition strongly increases chromosomal segregation errors and cell death and therefore, constitutes an efficient strategy for selectively eliminating tumor cells.

MPS1 inhibition in combination with microtubule-interfering agents is expected to improve therapeutic efficacy of anti-mitotic drugs and to overcome paclitaxel resistance.

The primary objectives of this study are to:

* Determine the safety, tolerability, maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of oral BAY1217389 given in combination with intravenous (IV) paclitaxel using an intermittent dosing schedule (2 days on / 5 days off) in subjects with advanced malignancies.
* Characterize the pharmacokinetics (PK) of oral BAY1217389 and IV paclitaxel.

The exploratory objectives of this study are to:

* Determine any preliminary clinical efficacy of oral BAY1217389 given in combination with IV paclitaxel compared to paclitaxel given alone.
* Determine pharmacodynamic (PD) target modulation effects (decrease in phosphorylated kinetochore-associated protein pKNL1 and potentially other biomarkers like activation of the p53 system) of oral BAY1217389 in mandatory paired fresh tumor biopsies (or in mandatory paired fresh skin punch biopsies depending on the status of the subject and the accessibility of the tumor) taken on Day 2 of Cycle 1 (C1D2) and on C1D3.
* Evaluate the effect of oral BAY1217389 on the activation of p53 in blood samples as PD biomarker (blood samples will be taken as a mandatory procedure to monitor PD effects on C1D 4, C1D 3, and C1D 2).
* Evaluate the effect of BAY1217389 on levels of tumor-derived free circulating deoxyribonucleic acid (DNA) in blood samples taken before the first dose of study treatment and on C1D3, C1D8, and C1D15

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >/= 18 years.
* Study population:

  * For the dose-escalation cohorts: Subjects with histologically or cytologically confirmed advanced malignancies (solid tumors), refractory to any standard therapy, have no standard therapy available
  * For the expansion cohort: Subjects with advanced, histologically or cytologically confirmed triple-negative breast cancer (TNBC), refractory to any standard therapy, have no standard therapy available, or subjects actively refused any standard treatment and / or if, in the judgment of the investigator, experimental treatment is clinically acceptable.
* Subjects must have evaluable or measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver, and renal functions.

Exclusion Criteria:

* Known hypersensitivity to the study drugs or excipients of the preparations or any agent given in association with this study.
* Evidence of peripheral neuropathy of Grade >2.
* History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class >II, unstable angina (anginal symptoms at rest), new-onset angina (within the past 3 months before study entry), myocardial infarction within the past 3 months before study entry, or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers, calcium channel blockers, and digoxin are permitted).
* Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg, despite optimal medical management.
* Moderate or severe hepatic impairment, i.e. Child-Pugh class B or C.
* History of human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 28 days (Cycle 1)
  The MTD is defined as the highest dose that can be given such that the dose-limiting toxicity (DLT) rate of the combination treatment is not more than 10% higher than the cumulative DLT rate of the standard single-agent treatment across all previous and the current cohort.
Number of subjects with adverse events and serious adverse events as a measure of safety and tolerability. | After the first study drug administration and up to 30 days after the end of treatment with study drug before primary completion analysis of the study, up to 3 years
Maximum observed drug concentration (Cmax) of BAY1217389 in plasma | From pre-dose up to 96 hours post-dose on C1D-8 and C1D-4; from pre-dose up to 12 hours post-dose on C1D8 and C1D9
Area under the concentration versus time curve from zero to 12 hours (AUC [0-12]) of BAY1217389 in plasma | From pre-dose up to 12 hours post-dose on C1D-4, C1D8 and C1D9
Area under the concentration versus time curve from zero to 96 hours (AUC [0-96]) of BAY1217389 in plasma | From pre-dose up to 96 hours post-dose on C1D-4
Maximum observed drug concentration (Cmax) of paclitaxel in plasma | From pre-dose up to 24 hours post-dose on C1D1 and C1D8
Area under the concentration versus time curve from zero to infinity (AUC) of paclitaxel in plasma | From pre-dose up to 24 hours post-dose on C1D1 and C1D8

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (6):
  - Santa Monica, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Hackensack, New Jersey
  - Houston, Texas
  - San Antonio, Texas
- Rotterdam, Netherlands